CLINICAL TRIAL: NCT03637062
Title: Verify the Safety and Effectiveness of the Cerclage Pessary in the Prevention and Treatment of High-risk Preterm Pregnancy
Brief Title: Verify the Safety and Effectiveness of the Cerclage Pessary in Prevention and Treatment of High-risk Preterm Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: QH Medical Technology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QH-20170928
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: High Risk Pregnancy
MeSH Terms: interventions — Progesterone; Utrogestan; Pessaries

STUDY DESIGN:
Intervention Model Description: Open Multicentre Randomized Controlled Trial, in parallel groups, based on treatment with progesterone comparing the placement of a prophylactic cervical pessary with usual management in singleton pregnancies at high-risk of PTB due to a history of at least one previous preterm delivery and/or a history of late abortion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pessary (Experimental): the test group is pessary.The pregnant woman is assigned to the pessary group and after having excluded a vaginal infection the pessary will be inserted directly.
  Interventions: Device: pessary
- Progesterone (Active Comparator): the control group is progesterone. Pregnant women in the control group were treated by 200 mg QN, it is used for 34 gestational weeks.
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — progeaterone:Utrogestan is one of the normal drugs in China to prevent spontaneous preterm birth, the Utrogestan used in this study is from Laboratories Besins International.
  Other Names: Utrogestan
  Arms: Progesterone
Device: pessary — pessary: The cervical pessary is a vaginal device (silicone ring) that is used to treat pregnant women for preventing spontaneous preterm birth.
  Arms: pessary

SUMMARY:
Verify the safety and effectiveness of the cerclage pessary in the prevention and treatment of high-risk preterm pregnancy.

DETAILED DESCRIPTION:
Prospective Open-label Multicentre Randomized Controlled Trial. high-risk preterm pregnancy is that there are at least one history of spontaneous preterm birth and/or late abortion before 34+0 weeks, for high-risk pregnant women that meet the inclusion criteria, the early treatment with cerclage pessary at 12-18weeks compare with routine treatment. The patients will be informed of the intended therapeutic effect and possible side effects. If they agree and after obtaining their informed consent, they will be randomized to test group (cerclage pessary group) and control group (Utrogestan group).

ELIGIBILITY:
Inclusion Criteria:

* Women with a pregnancy and a history of at least one spontaneous preterm birth before 34+0 weeks and/or a history of late abortion
* 12+0 -18+0 weeks of gestation
* Minimal age of 18 years
* Informed consent signature

Exclusion Criteria:

* The previous preterm delivery is iatrogenic proterm labor
* Major fetal abnormalities (requiring surgery or leading to infant death or severe handicap)
* The pregnant woman with severe cervical erosion, cervical polyp, hemorrhage and the doctors think she could not use cerclage pessary
* The pregnant woman with uterine cervicitis
* The pregnant woman that has been confirmed premature birth
* Cerclage prior to randomisation
* Cerclage prior to randomisation
* Placenta previa totalis
* Active vaginal bleeding at the moment of randomization
* Spontaneous rupture of membranes at the time of randomization
* Silicone allergy
* Painful regular uterine contractions
* The pregnant woman have the indication of operation cervical cerclage
* Current participation in other RCT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Child's birth and survival（rate） | 34+0 weeks
  Child's birth and survival

SECONDARY OUTCOMES:
Time to birth of Offspring（gestational weeks） | before 37+0 weeks
  * Preterm birth before 37 weeks: rate of delivery before 36+6 weeks
  * Preterm birth before 34 weeks: rate of delivery before 33+6 weeks
  * Preterm birth before 32 weeks: rate of delivery before 31+6 weeks
  * Preterm birth before 30 weeks: rate of delivery before 29+6 weeks
  * Preterm birth before 28 weeks: rate of delivery before 27+6 weeks
Birth weight of Offspring(g) | before 37+0 weeks
  median weight (g) of the newborns at birth
Fetal or neonatal death （rate） | before 37+0 weeks
  rate of intrauterine demise or neonatal death during the first 24 hours
Neonatal morbidity （rate） | before 37+0 weeks
  rate of major adverse neonatal outcomes before discharge from the hospital：
  * Intraventricular Haemorrhage (IVH): grades III-IV
  * Retinopathy of prematurity
  * Respiratory Distress Syndrome (RDS): grades II-IV
  * Need for ventilation > 72 h
  * Necrotising enterocolitis
  * Proven or suspected sepsis, antibiotics (>5 days)
  * Need (Duration in days) for neonatal special care (NICU)
Harm from intervention（Case Report Form） | before 37+0 weeks
  Harm from intervention
Maternal death（rate） | before 37+0 weeks
  Maternal death
Significant maternal adverse events (rate) | before 37+0 weeks
  * Heavy bleeding: bleeding that requires a medical intervention
  * Cervical tear: cervical rupture due to the pessary placement
  * Uterine rupture: rupture of the uterus due to contractions or surgery
Physical or psychological intolerance to pessary for mother(number of cases) | before 37+0 weeks
  discomfort or pain due to the pessary that makes daily life uncomfortable
Rupture of membranes before 32 weeks for mother（rate） | before 37+0 weeks
  rate of rupture of amniotic membranes before 31+6 weeks
inflammation 3rd stage of chorioamnionitis（rate） | before 37+0 weeks
  inflammation 3rd stage of chorioamnionitis
Hospitalisation for threatened preterm labour before 32 weeks（Case Report Form） | before 37+0 weeks
  requirement of hospitalisation due to preterm contractions that need medical treatment to try to stop them before 31+6 weeks
  * Mean hospital stay duration: number of days of admittance at the hospital
  * Use of tocolytic treatment: Type of tocolytic, days of treatment, dose

REFERENCES:
- [Derived] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA, Aboelfadle Mohamed A. Cervical pessary for preventing preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2022 Dec 1;12(12):CD014508. doi: 10.1002/14651858.CD014508. PMID 36453699

DOCUMENTS (1):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT03637062/Prot_000.pdf